CLINICAL TRIAL: NCT07278895
Title: A Randomized Prospective Trial Comparing Dural Puncture Epidural (DPE) and Standard Epidural Analgesia for Labor in Term Pregnant Women"
Brief Title: Dural Puncture Epidural vs Standard Epidural Analgesia in Labor
Acronym: DPE-LABOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Baran, Clinical Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 423
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related; Analgesia, Epidural; Labor Pain
Keywords: Dural Puncture Epidural; Standard Epidural Analgesia; Labor Analgesia
MeSH Terms: conditions — Agnosia; Labor Pain

STUDY DESIGN:
Intervention Model Description: This study uses a two-arm parallel assignment model in which eligible laboring women are randomized equally to receive either Dural Puncture Epidural (DPE) analgesia or Standard Epidural Analgesia. Both groups are managed and observed concurrently without crossover between interventions.
Masking Description: This is an open-label study. Due to the nature of the neuraxial procedures, the anesthesiologist performing the block cannot be blinded to the intervention. Participants and clinical staff are also aware of the assigned technique. No masking was applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dural Puncture Epidural (DPE) (Experimental): Participants receive Dural Puncture Epidural analgesia using a 27G Whitacre spinal needle inserted through the Tuohy needle before epidural catheter placement, without intrathecal drug administration.
  Interventions: Procedure: Dural Puncture Epidural (DPE)
- Standard Epidural Analgesia (Active Comparator): Participants in this arm receive Standard Epidural Analgesia. The epidural block is performed using a Tuohy needle without dural puncture, and an epidural catheter is inserted into the epidural space. After a negative test dose, a bolus of 10 mL 0.125% bupivacaine with 1.5 µg/mL fentanyl is administered.
  Interventions: Procedure: Standard Epidural Analgesia

INTERVENTIONS:
Procedure: Dural Puncture Epidural (DPE) — The Dural Puncture Epidural (DPE) technique is performed by inserting a 27-gauge Whitacre spinal needle through the Tuohy epidural needle to puncture the dura without intrathecal drug injection. After removal of the spinal needle, an epidural catheter is placed, and following a negative test dose, a bolus of 10 mL 0.125% bupivacaine with 1.5 µg/mL fentanyl is administered.
  Arms: Dural Puncture Epidural (DPE)
Procedure: Standard Epidural Analgesia — Standard Epidural Analgesia is performed using a Tuohy needle without dural puncture. An epidural catheter is inserted into the epidural space, and after a negative test dose, a bolus of 10 mL 0.125% bupivacaine with 1.5 µg/mL fentanyl is administered.
  Arms: Standard Epidural Analgesia

SUMMARY:
This randomized prospective study compares Dural Puncture Epidural (DPE) and Standard Epidural Analgesia in term laboring women. The study evaluates analgesic quality, onset time, maternal and neonatal outcomes, side effects, and overall patient satisfaction.

DETAILED DESCRIPTION:
This prospective randomized clinical trial is designed to compare the efficacy and safety of Dural Puncture Epidural (DPE) analgesia with Standard Epidural Analgesia in term laboring women requesting neuraxial analgesia. The DPE technique involves performing a dural puncture with a 27-gauge Whitacre spinal needle through the Tuohy epidural needle before catheter placement, without administering any intrathecal medication. In both groups, a bolus of 10 mL 0.125% bupivacaine with 1.5 µg/mL fentanyl is administered following a negative epidural test dose.

The primary objective of the study is to determine whether DPE provides a faster onset and higher quality of labor analgesia compared with the conventional epidural technique. Secondary objectives include evaluating maternal hemodynamic changes, sensory and motor block characteristics, the need for additional bolus doses, total local anesthetic consumption, maternal side effects (hypotension, nausea, vomiting, pruritus, urinary retention), post-dural puncture headache, fetal heart rate changes, Apgar scores, duration of labor, and overall patient satisfaction.

Term pregnant women aged 18-45 years with cervical dilation ≥4 cm, effacement ≥50-60%, and baseline VAS ≥3 will be included. Exclusion criteria include hypertensive disorders of pregnancy, placental abnormalities, contraindications to neuraxial anesthesia, morbid obesity (BMI ≥40), drug allergy, opioid dependence, or accidental dural puncture with the epidural needle. Eligible participants will be randomly assigned to either the DPE group or the Standard Epidural group in a 1:1 ratio. All procedures will be performed at the Gazi Yaşargil Training and Research Hospital by anesthesiologists experienced in obstetric neuraxial techniques, and data will be collected by an independent observer not involved in the block procedure.

The study aims to contribute to the growing body of evidence on optimizing labor analgesia techniques by determining whether the DPE approach leads to improved analgesic effectiveness, greater maternal comfort, and stable maternal-fetal outcomes compared with standard epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Term pregnant women (≥37 weeks of gestation).
2. Requesting neuraxial labor analgesia.
3. Age between 18 and 45 years.
4. ASA physical status I-II.
5. Cervical dilation ≥ 4 cm at the time of enrollment.
6. Cervical effacement ≥ 50-60%.
7. Baseline pain score of VAS ≥ 3.
8. Ability to provide informed consent.

Exclusion Criteria:

1. Hypertensive disorders of pregnancy (gestational hypertension, preeclampsia, eclampsia).
2. Placental abnormalities (placenta previa, placental abruption, etc.).
3. Contraindications to neuraxial anesthesia (coagulopathy, infection at puncture site, severe hypovolemia).
4. Known allergy or hypersensitivity to local anesthetics or opioids used in the study.
5. Morbid obesity (Body Mass Index ≥ 40 kg/m²).
6. Opioid dependence or chronic opioid use.
7. Accidental dural puncture with the epidural needle prior to randomization.
8. Multiple gestation or non-cephalic presentation (if clinically relevant to your protocol).
9. Fetal distress at the time of enrollment.
10. Patient refusal to participate.
11. Any condition deemed by the investigator to pose increased risk or interfere with study outcomes.

    -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligible participants are exclusively female due to the nature of the study, which involves labor analgesia in term pregnant women.
Enrollment: 102 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Time to Onset of Effective Analgesia (VAS < 3) | Within 30 minutes after epidural bolus
  Time in minutes from the administration of the initial epidural bolus until the patient reports a pain score of VAS < 3, indicating effective labor analgesia.

SECONDARY OUTCOMES:
Sensory Block Level | Within 30 minutes after epidural bolus
  The highest dermatome level of sensory block assessed by pinprick or cold test.
Motor Block Score (Bromage Score) | Within 30 minutes after epidural bolus
  Degree of motor block measured using the Bromage scale (0-3).
Need for Additional Epidural Bolus | During labor until delivery
  Number of additional boluses required when VAS ≥ 4.
Time to First Additional Bolus | From initiation of analgesia to delivery
  Total amount (mL) of local anesthetic administered during labor.
Maternal Hemodynamic Changes | First 30 minutes after epidural bolus
  Changes in systolic/diastolic blood pressure and heart rate compared to baseline
Maternal Side Effects | During labor until delivery
  Incidence of hypotension, nausea, vomiting, pruritus, urinary retention, or other complications.
Post-Dural Puncture Headache (PDPH) | Day 3 and Day 7 postpartum
  Presence or absence of typical post-dural puncture headache symptoms.
Fetal Heart Rate Changes | During labor until delivery
  Any abnormal fetal heart rate patterns following neuraxial analgesia.
Duration of Labor | From initiation of analgesia to delivery
  Time in minutes or hours from epidural bolus administration to birth.
Neonatal Apgar Scores | At 1 minute and 5 minutes after birth
  Neonatal Apgar scores assessed at 1 and 5 minutes postpartum.
Maternal Satisfaction Score | Immediately after delivery
  Patient satisfaction with labor analgesia measured on a 0-10 Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with qualified researchers upon reasonable request. Data will be provided via email after review and approval of the research proposal by the principal investigator.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available starting 6 months after publication of the study results and will remain available for up to 5 years.
Access Criteria: De-identified IPD will be shared via email upon reasonable request and PI approval.
  e-mail:mehmetbaran1492@gmail.com

REFERENCES:
- [Background] Pazur I, Ozegic O, Lijovic L, Jaic KK, Pesic M. The Efficacy of Dural Puncture Epidural Performed by 27-gauge Whitacre Needle in Labour Epidural Analgesia: Randomized Single-Blinded Controlled Study. Turk J Anaesthesiol Reanim. 2023 Aug 18;51(4):304-310. doi: 10.4274/TJAR.2023.221085. PMID 37587657